CLINICAL TRIAL: NCT05951699
Title: Prospective Clinical Trial to Assess a Mini-invasive Pre-surgical Procedure to Detect Residual Breast or Axillary Disease in Patients With cT1-T2-T3 cN0/N1 Breast Cancer in Complete Clinical/Radiological Remission After Primary Chemotherapy
Brief Title: Mini-invasive Detection of Residual Disease in Breast Cancer Patients in Remission After Primary Chemotherapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Other Study IDs: INT 198/21
Record Dates: First submitted 2023-06-01; First posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Neoadjuvant chemotherapy; vacuum-assisted biopsy
MeSH Terms: conditions — Breast Neoplasms | interventions — Biopsy, Needle

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- minimally invasive preoperative image-guided vacuum-assisted biopsy: cT1-cT2-cT3 cN0-cN1 breast cancer patients, either with clinical/radiological complete response, or with <1 cm residual breast disease after systemic primary treatment, undergo preoperative image-guided breast VAB with 9-gauge needle.
  Patients who are cN1 before systemic primary treatment undergo removal of the tagged axillary nodes.
  In both cases the aim is to identify any residual disease. Conservative breast surgery or mastectomy will be performed in all patients after multidisciplinary clinical evaluation.
  Surgically confirmed residual tumor will be compared to VAB result.
  Interventions: Device: minimally invasive preoperative image-guided vacuum-assisted biopsy

INTERVENTIONS:
Device: minimally invasive preoperative image-guided vacuum-assisted biopsy — minimally invasive preoperative image-guided vacuum-assisted biopsy of the breast and needle biopsy of axillary lymph node
  Other Names: needle biopsy

SUMMARY:
Breast surgery may be overtreatment when there is a complete response to systemic neoadjuvant treatment as determined clinically and by imaging. However the reliability of imaging techniques (ultrasound, mammography and magnetic resonance) in identifying complete response varies in published studies and surgery remains the preferred method of detecting residual disease.

The aims of this study are:

1. To assess the reliability of minimally invasive preoperative image-guided vacuum-assisted biopsy (VAB) in identifying residual breast in cT1-cT2-cT3, cN0-cN1 breast cancer patients, either with complete clinical/radiological response, or with residual breast disease <1 cm, after systemic neoadjuvant treatment.
2. To assess the reliability of minimally invasive preoperative image-guided needle biopsy in identifying residual axillary disease in cT1-cT2-cT3, cN0-cN1 breast cancer patients, either with complete clinical/radiological response, or with residual breast disease <1 cm, after systemic neoadjuvant treatment.

After neoadjuvant treatment, and evaluation with ultrasound, mammography and magnetic resonance, VAB will be performed on the breast, and needle biopsy will be performed on the axillary lymph node of pre-treatment cN1 cases, previously marked with a magnetic clip.

The biopsy findings will be compared with the surgical findings, consisting in quadrantectomy or mastectomy plus sentinel node biopsy (or separate removal of tagged lymph nodes if they do not coincide with the sentinel node(s)) to assess the ability of biopsy to identify residual disease.

DETAILED DESCRIPTION:
Systemic neoadjuvant treatment was introduced in the 1990s (1,2) mainly for advanced (cT2, cT3) breast cancer to reduce the extent of disease and hence allow conservative surgery instead of mastectomy.

Studies (3-6) demonstrated that pathologic complete response (pCR) in the breast and/or axilla after neoadjuvant treatment predicted better overall survival (OS), better distant relapse-free survival (DRS), and lower mortality.

More recently, targeted neoadjuvant therapies achieve pCR in over 60% of patients (7,8) and in up to 70% of patients with HER2-positive or triple negative subtypes that are generally associated with poorer outcomes (9).

Ultrasound, mammography and magnetic resonance imaging are still imprecise in identifying surgically confirmed residual disease after neoadjuvant chemotherapy (10,11) and the sensitivity and specificity of these imaging techniques vary markedly, (12) so surgery remains the most reliable method of detecting any residual disease.

The aims of this study are

1. to evaluate the ability of minimally invasive preoperative image-guided vacuum-assisted biopsy (VAB) to identify residual breast disease in breast cancer patients with either complete clinical/radiological complete response or with residual disease <1 cm after systemic neoadjuvant treatment; and
2. to evaluate the ability of biopsy to identify residual axillary lymph node disease in patients who are cN1 pre-treatment and whose suspicious nodes are marked with a metal clip before treatment.

The VAB/needle biopsy results will be compared to pathological findings after quadrantectomy/mastectomy or surgical removal of the sentinel axillary lymph node(s) and tagged axillary lymph node(s) (if distinct from the sentinel node(s)).

This study is being conducted with a view to performing a future clinical trial on the omission of surgery in cases with clinical/radiological complete response and negative preoperative VAB.

ELIGIBILITY:
Inclusion Criteria:

* Radiologically confirmed unifocal cT1-cT2-cT3 cN0-cN1 breast cancer patients indicated for primary chemotherapy
* Histologically confirmed HER2-positive, triple negative or luminal B HER2-positive invasive breast cancer
* Clinical/radiological complete response or residual breast disease <1 cm after primary chemotherapy
* Absence of locoregional relapse or distant metastasis
* Signed informed consent to participate.

Exclusion Criteria:

* Disease surgically inoperable or surgery not performed
* Multifocal disease or presence of microcalcifications at imaging.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: cT1-cT2-cT3 cN0-cN1 breast cancer patients, either with clinical/radiological complete response, or with <1 cm residual breast disease after systemic primary treatment
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2022-04-28 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the accuracy of histological examination of the breast VAB performed pre-surgery | 40 days
  Identification of percentage of cases with correspondence between pre-operative VAB findings in breast with histological findings after quadrantectomy or mastectomy in patients with complete radiological response after neoadjuvant chemotherapy.

SECONDARY OUTCOMES:
Evaluation of the accuracy of histological examination of the lymph node biopsy performed pre-surgery | 40 days
  Identification of percentage of cases with correspondence between pre-operative biopsy findings in tagged cN1 axillary lymph nodes with histological findings after sentinel node biopsy and surgical removal of the tagged node/s (if different from the sentinel node(s)).

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Martelli, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Via G. Venezian 1, 20133 Milan, Italy
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Bonadonna G, Veronesi U, Brambilla C, Ferrari L, Luini A, Greco M, Bartoli C, Coopmans de Yoldi G, Zucali R, Rilke F, et al. Primary chemotherapy to avoid mastectomy in tumors with diameters of three centimeters or more. J Natl Cancer Inst. 1990 Oct 3;82(19):1539-45. doi: 10.1093/jnci/82.19.1539. PMID 2402015
- [Result] Fisher B, Brown A, Mamounas E, Wieand S, Robidoux A, Margolese RG, Cruz AB Jr, Fisher ER, Wickerham DL, Wolmark N, DeCillis A, Hoehn JL, Lees AW, Dimitrov NV. Effect of preoperative chemotherapy on local-regional disease in women with operable breast cancer: findings from National Surgical Adjuvant Breast and Bowel Project B-18. J Clin Oncol. 1997 Jul;15(7):2483-93. doi: 10.1200/JCO.1997.15.7.2483. PMID 9215816
- [Result] Esserman LJ, Berry DA, DeMichele A, Carey L, Davis SE, Buxton M, Hudis C, Gray JW, Perou C, Yau C, Livasy C, Krontiras H, Montgomery L, Tripathy D, Lehman C, Liu MC, Olopade OI, Rugo HS, Carpenter JT, Dressler L, Chhieng D, Singh B, Mies C, Rabban J, Chen YY, Giri D, van 't Veer L, Hylton N. Pathologic complete response predicts recurrence-free survival more effectively by cancer subset: results from the I-SPY 1 TRIAL--CALGB 150007/150012, ACRIN 6657. J Clin Oncol. 2012 Sep 10;30(26):3242-9. doi: 10.1200/JCO.2011.39.2779. Epub 2012 May 29. PMID 22649152
- [Result] Shin HC, Han W, Moon HG, Im SA, Moon WK, Park IA, Park SJ, Noh DY. Breast-conserving surgery after tumor downstaging by neoadjuvant chemotherapy is oncologically safe for stage III breast cancer patients. Ann Surg Oncol. 2013 Aug;20(8):2582-9. doi: 10.1245/s10434-013-2909-6. Epub 2013 Mar 16. PMID 23504119
- [Result] von Minckwitz G, Untch M, Blohmer JU, Costa SD, Eidtmann H, Fasching PA, Gerber B, Eiermann W, Hilfrich J, Huober J, Jackisch C, Kaufmann M, Konecny GE, Denkert C, Nekljudova V, Mehta K, Loibl S. Definition and impact of pathologic complete response on prognosis after neoadjuvant chemotherapy in various intrinsic breast cancer subtypes. J Clin Oncol. 2012 May 20;30(15):1796-804. doi: 10.1200/JCO.2011.38.8595. Epub 2012 Apr 16. PMID 22508812
- [Result] Martelli G, Miceli R, Folli S, Guzzetti E, Chifu C, Maugeri I, Ferranti C, Bianchi G, Capri G, Carcangiu ML, Paolini B, Agresti R, Ferraris C, Piromalli D, Greco M. Sentinel node biopsy after primary chemotherapy in cT2 N0/1 breast cancer patients: Long-term results of a retrospective study. Eur J Surg Oncol. 2017 Nov;43(11):2012-2020. doi: 10.1016/j.ejso.2017.07.023. Epub 2017 Aug 10. PMID 28912071
- [Result] Haque W, Verma V, Hatch S, Suzanne Klimberg V, Brian Butler E, Teh BS. Response rates and pathologic complete response by breast cancer molecular subtype following neoadjuvant chemotherapy. Breast Cancer Res Treat. 2018 Aug;170(3):559-567. doi: 10.1007/s10549-018-4801-3. Epub 2018 Apr 24. PMID 29693228
- [Result] Goorts B, van Nijnatten TJ, de Munck L, Moossdorff M, Heuts EM, de Boer M, Lobbes MB, Smidt ML. Clinical tumor stage is the most important predictor of pathological complete response rate after neoadjuvant chemotherapy in breast cancer patients. Breast Cancer Res Treat. 2017 May;163(1):83-91. doi: 10.1007/s10549-017-4155-2. Epub 2017 Feb 15. PMID 28205044
- [Result] Santonja A, Sanchez-Munoz A, Lluch A, Chica-Parrado MR, Albanell J, Chacon JI, Antolin S, Jerez JM, de la Haba J, de Luque V, Fernandez-De Sousa CE, Vicioso L, Plata Y, Ramirez-Tortosa CL, Alvarez M, Llacer C, Zarcos-Pedrinaci I, Carrasco E, Caballero R, Martin M, Alba E. Triple negative breast cancer subtypes and pathologic complete response rate to neoadjuvant chemotherapy. Oncotarget. 2018 May 29;9(41):26406-26416. doi: 10.18632/oncotarget.25413. eCollection 2018 May 29. PMID 29899867
- [Result] Chagpar AB, Middleton LP, Sahin AA, Dempsey P, Buzdar AU, Mirza AN, Ames FC, Babiera GV, Feig BW, Hunt KK, Kuerer HM, Meric-Bernstam F, Ross MI, Singletary SE. Accuracy of physical examination, ultrasonography, and mammography in predicting residual pathologic tumor size in patients treated with neoadjuvant chemotherapy. Ann Surg. 2006 Feb;243(2):257-64. doi: 10.1097/01.sla.0000197714.14318.6f. PMID 16432360
- [Result] Croshaw R, Shapiro-Wright H, Svensson E, Erb K, Julian T. Accuracy of clinical examination, digital mammogram, ultrasound, and MRI in determining postneoadjuvant pathologic tumor response in operable breast cancer patients. Ann Surg Oncol. 2011 Oct;18(11):3160-3. doi: 10.1245/s10434-011-1919-5. Epub 2011 Sep 27. PMID 21947594
- [Result] Fowler AM, Mankoff DA, Joe BN. Imaging Neoadjuvant Therapy Response in Breast Cancer. Radiology. 2017 Nov;285(2):358-375. doi: 10.1148/radiol.2017170180. PMID 29045232
- [Result] Heil J, Pfob A, Sinn HP, Rauch G, Bach P, Thomas B, Schaefgen B, Kuemmel S, Reimer T, Hahn M, Thill M, Blohmer JU, Hackmann J, Malter W, Bekes I, Friedrichs K, Wojcinski S, Joos S, Paepke S, Ditsch N, Rody A, Grosse R, van Mackelenbergh M, Reinisch M, Karsten M, Golatta M; RESPONDER Investigators. Diagnosing Pathologic Complete Response in the Breast After Neoadjuvant Systemic Treatment of Breast Cancer Patients by Minimal Invasive Biopsy: Oral Presentation at the San Antonio Breast Cancer Symposium on Friday, December 13, 2019, Program Number GS5-03. Ann Surg. 2022 Mar 1;275(3):576-581. doi: 10.1097/SLA.0000000000004246. PMID 32657944
- [Result] Buderer NM. Statistical methodology: I. Incorporating the prevalence of disease into the sample size calculation for sensitivity and specificity. Acad Emerg Med. 1996 Sep;3(9):895-900. doi: 10.1111/j.1553-2712.1996.tb03538.x. PMID 8870764